CLINICAL TRIAL: NCT06607952
Title: Experiential Learning and Critical Thinking: An Exploration of the Learning Effectiveness of Using Situational Case Videos in the Application of Emergency Nursing Course
Acronym: Non
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Chia-Chi Kuo, Associate Professor, Chang Gung University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202400142B0; EZRPF6P0041 (Other Grant/Funding Number: MOE teaching practice research program of Taiwan)
Record Dates: First submitted 2024-09-14; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Nursing Students With no Specific Health Issues
Keywords: emergency nursing; nursing students; scenario-based case videos; experiential learning; critical thinking

STUDY DESIGN:
Intervention Model Description: This study is a two-group, pre- and post-test, parallel, non-blind randomized controlled trial. Participants will be randomly assigned to either the experimental group class or the control group class.
Masking Description: Non
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group with scenario-based case videos teaching method. (Experimental): The students in the experimental group will receive a new teaching method of five scenario-based case videos. These scenarios include Triage, SDH (Subdural Hemorrhage) and ETTC (Emergency Trauma Training Course), AMI (Acute Myocardial Infarction) and D2B (Door to Balloon), COPD AE (Chronic Obstructive Pulmonary Disease with Acute Exacerbation) and TOCC (Travel, Occupation, Contact, and Cluster History Review), and Sepsis and CVC Procedure (Central Venous Catheter Procedure).
  Interventions: Other: scenario-based case videos teaching protocol
- The control group with traditional lecture-based teaching method. (Active Comparator): The students in the control group will receive traditional lecture-based teaching on the five topics: Triage, SDH and ETTC, AMI and D2B, COPD AE and TOCC, and Sepsis and CVC Procedure.
  Interventions: Other: traditional lecture-based teaching method

INTERVENTIONS:
Other: scenario-based case videos teaching protocol — Students in the experimental group will receive a new teaching method of scenario-based case video interventions. These videos cover five key scenarios: Triage, SDH and ETTC, AMI and D2B, COPD AE and TOCC, and Sepsis and the CVC Procedure.
  This teaching method is grounded in experiential learning theory and critical thinking strategies, designed to guide students in learning emergency nursing through video experiences. In each class, the instructor will first introduce the foundational concepts of emergency nursing for each system. Students will then watch a 15-minute scenario-based case video. Afterward, the instructor will facilitate a 15-minute discussion using reflection sheets to promote experiential learning and critical
  Arms: The experimental group with scenario-based case videos teaching method.
Other: traditional lecture-based teaching method — Students in the control group will receive traditional lecture-based instruction on the five topics: Triage, SDH and ETTC , AMI and D2B , COPD AE and TOCC , and Sepsis and the CVC Procedure. During the lectures, the instructor will encourage students to ask questions and engage in discussions to enhance understanding.
  Arms: The control group with traditional lecture-based teaching method.

SUMMARY:
This study is a randomized controlled trial. The goal of this clinical trial is to introduce scenario-based case videos into the elective course of Emergency Nursing and Applications for first-year students in a two-year program. By using five typical scenario-based case videos, the aim is to guide students through experiential learning and critical thinking, overcome learning difficulties, increase learning interest, and enhance learning outcomes.

The main aims of this research are:

To explore the effectiveness of emergency scenario-based case teaching on students learning focus, knowledge acquisition, classroom participation, and course satisfaction

The main questions it aims to answer are:

1. Are there significant differences in emergency nursing knowledge, learning focus, and course satisfaction between students in the experimental group and the control group after different teaching methods are applied?
2. Are there significant differences in classroom participation rates and attendance rates between students in the experimental group and the control group under different teaching methods?

DETAILED DESCRIPTION:
This study is a two-group, pre- and post-test, parallel, non-blind randomized controlled trial. This educational practice research project will use scenario-based case videos as the intervention, with experiential learning and critical thinking as the teaching strategies. The goal is to guide students through experiential learning of emergency nursing via videos, using the seven core competencies of the mini-CEX (Physical Assessment, Clinical Judgment, Nursing Interventions, Communication, Empathy, Counseling and Education, Teamwork) to design lesson plans, reflection sheets, and learning materials. Students will be encouraged to critical thinking health issues, strengths, weaknesses, and improvement suggestions in the care process, providing feedback on emergency care.

This study will design five scenario-based lesson plans on topics including triage, meningeal hemorrhage, acute myocardial infarction, acute exacerbation of chronic obstructive pulmonary disease, and sepsis. Videos for these scenarios will be created and edited based on these lesson plans.

Convenience sampling will be used to select first-year nursing students from a technology university in Southern Taiwan as participants. Classes will be randomly assigned to either the experimental group or the control group, with an estimated sample size of about 50-60 students per class, totaling 120 participants.

The experimental group will receive the new teaching method involving five scenario-based case videos, while the control group will continue with the traditional lecture-based method. Both groups will complete a basic information questionnaire and a pre-test of prior knowledge. At the end of the semester, students will undergo a post-test assessing emergency nursing knowledge, learning focus, and course satisfaction. Teachers will calculate the overall classroom participation rate, attendance rate, and perform a qualitative analysis of learning materials and reflective reports from the experimental group.

The researcher will screen and recruit subjects, conduct the intervention, and collect data. Inferential statistics will be performed using chi-square tests, Fisher's Exact Test, and independent t-tests to compare differences in basic attributes, knowledge, learning focus, course satisfaction, classroom participation rates, and attendance rates between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* First-year students in the two-year nursing program at a technology university in Southern Taiwan.
* Adults aged 18 and above.
* Enrolled in the elective course "Emergency Nursing and Applications."

Exclusion Criteria:

* Students who have not previously completed courses in Anatomy and Physiology, Basic Nursing, Medical-Surgical Nursing, Physical Assessment, or Pharmacology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-03 (Estimated); Primary Completion 2025-01-09 (Estimated); Study Completion 2025-01-09 (Estimated)

PRIMARY OUTCOMES:
Emergency Nursing Knowledge Test | post-lesson quizzes after the course and a final exam at the end of the semester (through study completion, an average of 4.5 months).
  Emergency Nursing Knowledge Test: covering four units: subdural hemorrhage, acute myocardial infarction, acute exacerbation of chronic obstructive pulmonary disease, and sepsis. An average of 20 single-choice questions, with a total score ranging from 0 to 100, where higher scores indicate a greater knowledge of Emergency Nursing.
Learning Worksheets | during the course on week 1, 4, 6, 10, 14.
  Learning Worksheets: covering five units-triage, subdural hemorrhage, acute myocardial infarction, acute exacerbation of chronic obstructive pulmonary disease, and sepsis. Each unit has 10 fill-in-the-blank questions, with a total score ranging from 0 to 100, where higher scores indicate a greater learning efficacy.
Learning Engagement Scale | through study completion (at the end of the semester), an average of 4.5 months.
  Learning Engagement Scale: The scale consists of 19 single-choice questions scored using a five-point Likert scale, ranging from 1 to 5. The higher scores indicating greater classroom engagement. The internal consistency (Cronbach's α) of the original scale ranges from 0.83 to 0.88.
Course Satisfaction Questionnaire | through study completion (at the end of the semester), an average of 4.5 months.
  Course Satisfaction Questionnaire: The questionnaire consists of 12 items, rated on a five-point Likert scale, where 1 indicates strong disagreement and 5 indicates strong agreement. Higher scores indicate higher student satisfaction with the course.

SECONDARY OUTCOMES:
Class Discussion Participation Rate | through study completion (at the end of the semester), an average of 4.5 months.
  Class Discussion Participation Rate: The discussion participation rate for each teaching unit = (Number of students participating in the discussion ÷ Total number of students in the class) × 100%.
Class Attendance Rate | through study completion (at the end of the semester), an average of 4.5 months.
  The attendance rate for each teaching unit = (Number of students present ÷ Total number of students in the class) × 100%.

OTHER OUTCOMES:
Prior Knowledge Test | Baseline (Before intervention (at the start of the semester)).
  Prior Knowledge Test: This study developed a prior knowledge test based on the essential knowledge required for emergency nursing, including topics such as anatomy and physiology, basic nursing, medical-surgical nursing, and physical assessment. Total 20 single-choice questions, with a total score ranging from 0 to 100, where higher scores indicate a greater prior knowledge of Emergency Nursing.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University of Science and Technology, Chiayi Campus, Chiayi City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
We will not to share individual participant data due to school policy.

REFERENCES:
- See also: Related Info — https://doi.org/10.26355/eurrev_202104_25726